CLINICAL TRIAL: NCT06329700
Title: Performance of Parenchymal Sparing Hepatectomy in Patients With CLM and Post-chemotherapy Liver Atrophy
Brief Title: Parenchymal Sparing Hepatectomy in Post-chemotherapy Liver Atrophy
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Matteo Donadon, Professor of Surgery, Head Surgical Oncology Program, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: ParSparInLivAtrophy
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer Stage IV
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No post-chemotherapy liver atrophy: Patients treated with systemic chemotherapy, then hepatectomy for colorectal liver metastases. No occurrence of post-chemotherapy liver atrophy as measured by computed-tomography liver volumetry.
  Interventions: Procedure: Hepatectomy
- Yes post-chemotherapy liver atrophy: Patients treated with systemic chemotherapy, then hepatectomy for colorectal liver metastases. Yes, occurrence of post-chemotherapy liver atrophy as measured by computed-tomography liver volumetry.
  Interventions: Procedure: Hepatectomy

INTERVENTIONS:
Procedure: Hepatectomy — Surgical removal of a part of the liver
  Other Names: Liver resection

SUMMARY:
Major hepatectomy in patients with colorectal liver metastases (CLM) and post-chemotherapy liver atrophy is associated with increased complications. Whether the performance of parenchymal-sparing hepatectomy (PSH) in those patients can be safer is unknown. The aim of this study was to assess the clinical impact of post-chemotherapy liver atrophy on patients undergoing PSH for CLM. For this purpose, the occurrence of liver atrophy was recorded and then computed against the occurrence of postoperative morbidity and mortality.

DETAILED DESCRIPTION:
Patients affected by CLMs and trated with neoadjuvant systemic chemotherapy and then hepatectomy were reviewed with the intent to assess the occurrence of liver atrophy, which is a sign of liver dysfunction and a source of morbidity expecially in patients treated with major or extended hepatectomy. Whether the performance of parenchymal-sparing hepatectomy (PSH) in those patients can be safer is unknown. Then, we planned to review our cases with the above mentioned endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with multiple CLMs treated with preoperative chemotherapy and parenchymal sparing surgery;
* Only patients with available volumetry of the pre- and post-chemotherapy abdominal enhanced computed tomography (CT) images;

Exclusion Criteria:

* Patients who underwent preoperative PVE;
* Patients treated by major hepatectomies; Patients treated with thermal ablation alone or in association with hepatic resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by colorectal liver metastases awaiting liver surgery, and receiving before surgery systemic chemotherapy (neoadjuvant).
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | From the date of surgery up to 90 days
  Any adverse event after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Donadon, MD, PhD, Principal Investigator — University of Eastern Piedmont

IPD SHARING:
Plan to Share IPD: Yes
Yes, after reasonable request.
Supporting Information: Study Protocol
Time Frame: After pubblication of the paper(s). No limit in time.
Access Criteria: Reasonable request to the PI or corresponsing author.

REFERENCES:
- [Result] Yamashita S, Shindoh J, Mizuno T, Chun YS, Conrad C, Aloia TA, Vauthey JN. Hepatic atrophy following preoperative chemotherapy predicts hepatic insufficiency after resection of colorectal liver metastases. J Hepatol. 2017 Jul;67(1):56-64. doi: 10.1016/j.jhep.2017.01.031. Epub 2017 Feb 10. PMID 28192187
- [Result] Omichi K, Yamashita S, Cloyd JM, Shindoh J, Mizuno T, Chun YS, Conrad C, Aloia TA, Vauthey JN, Tzeng CD. Portal Vein Embolization Reduces Postoperative Hepatic Insufficiency Associated with Postchemotherapy Hepatic Atrophy. J Gastrointest Surg. 2018 Jan;22(1):60-67. doi: 10.1007/s11605-017-3467-1. Epub 2017 Jun 5. PMID 28585106
- [Result] Torzilli G, Procopio F, Botea F, Marconi M, Del Fabbro D, Donadon M, Palmisano A, Spinelli A, Montorsi M. One-stage ultrasonographically guided hepatectomy for multiple bilobar colorectal metastases: a feasible and effective alternative to the 2-stage approach. Surgery. 2009 Jul;146(1):60-71. doi: 10.1016/j.surg.2009.02.017. PMID 19541011
- [Result] Tani K, Shindoh J, Takamoto T, Shibahara J, Nishioka Y, Hashimoto T, Sakamoto Y, Hasegawa K, Makuuchi M, Kokudo N. Kinetic Changes in Liver Parenchyma After Preoperative Chemotherapy for Patients with Colorectal Liver Metastases. J Gastrointest Surg. 2017 May;21(5):813-821. doi: 10.1007/s11605-017-3359-4. Epub 2017 Jan 12. PMID 28083837